CLINICAL TRIAL: NCT03105271
Title: Acute Kidney Injury in Patients With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey D. Lebensburger, DO, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: AKISCD
Record Dates: First submitted 2017-03-23; First posted 2017-04-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Sickle Cell Disease; Kidney Injury; Kidney Diseases; Kidney Disease, Chronic
MeSH Terms: conditions — Anemia, Sickle Cell; Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and blood will be stored in biorepository.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with sickle cell disease may be at risk for acute kidney injury (AKI)during sickle cell crisis (pain or acute chest syndrome). This study will evaluate the role of hemolysis during SCD crisis on the development of AKI and the role for monitoring urine biomarkers during an admission for crisis and during well clinic follow-up.

DETAILED DESCRIPTION:
Patients admitted to the hospital for acute chest syndrome or vaso-occlusive pain events may consent to participate in this study. Patients will consent to daily blood and urine collection during their hospitalization and during well clinic visits.

Each AM, participants will have blood and urine collected, processed, and strored for future analysis of hemolytic markers and biomarkers of kidney injury. Patients will also have strict urine output recorded. Acute kidney injury (AKI) will be defined by the current KDIGO definition based on either a rise in serum creatinine or decline in urine output. Patient medical course will be reviewed to determine interventions and outcomes of their admission based on the development of AKI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HbSS or SB0 thalassemia admitted for vaso-occlusive pain crisis or acute chest syndrome
* Able to sign informed consent

Exclusion Criteria:

-

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with HbSS or SB0 thalassemia admitted to Children's of Alabama for a vaso-occlusive pain crisis or acute chest syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute Kidney Injury | Hospitalizations through study completion, an average of one year
  Evaluate the incidence of KDIGO defined AKI among patients admitted for pain or acute chest syndrome. AKI is defined by KDIGO as an increase in SCr by 50% or ≥0.3mg/dL from baseline, or UOP <0.5mL/kg/hr for 12 hrs
Impact of Acute Kidney Injury during Pain or Acute Chest Syndrome Hospitalizations on the Development of Chronic Kidney Disease as defined by KDIGO. | One year
  We will evaluate the impact of AKI on eGFR. To evaluate this impact, we will compare the change in eGFR, as measured by cystatin C, obtained from each patient during their non-acute clinic visit both immediately prior to their AKI events and after AKI events.
Impact of free heme and endothelin on development of AKI | two years
  We will test the hypothesis that free heme and endothelin are elevated in patients that develop AKI as compared to patients without AKI.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baddam S, Aban I, Hilliard L, Howard T, Askenazi D, Lebensburger JD. Acute kidney injury during a pediatric sickle cell vaso-occlusive pain crisis. Pediatr Nephrol. 2017 Aug;32(8):1451-1456. doi: 10.1007/s00467-017-3623-6. Epub 2017 Feb 25. PMID 28238158
- [Background] Lebensburger JD, Palabindela P, Howard TH, Feig DI, Aban I, Askenazi DJ. Prevalence of acute kidney injury during pediatric admissions for acute chest syndrome. Pediatr Nephrol. 2016 Aug;31(8):1363-8. doi: 10.1007/s00467-016-3370-0. Epub 2016 Mar 24. PMID 27011218
- [Background] Oakley J, Zahr R, Aban I, Kulkarni V, Patel RP, Hurwitz J, Askenazi D, Hankins J, Lebensburger J. Acute Kidney Injury during Parvovirus B19-Induced Transient Aplastic Crisis in Sickle Cell Disease. Am J Hematol. 2018 May 14:10.1002/ajh.25140. doi: 10.1002/ajh.25140. Online ahead of print. No abstract available. PMID 29756409